CLINICAL TRIAL: NCT05155410
Title: Effect of 14 Days of Exogenous Ketone Supplementation on Glycemic Control in Type 2 Diabetes: a Randomized Placebo-controlled Crossover Trial
Brief Title: Examining the Effect of Exogenous Ketone Supplementation on Glucose Control in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Associate professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: H21-01762
Record Dates: First submitted 2021-11-30; First posted 2021-12-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: 3-Hydroxybutyric Acid; Glycemic Control; Hyperglycemia; Ketones; Glucose Control; Inflammation; Immune cell function; Cognition
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hyperglycemia; Ketosis; Inflammation | interventions — Flavoring Agents

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Participants will consume 15 g of an active oral exogenous ketone monoester supplement 15 minutes prior to each meal of the day for a 14-day period.
  Pre-intervention (baseline) and post-intervention measurements will be obtained before and immediately after the 14-day period.
  All meals will be provided throughout the supplementation period Participants will wear a continuous glucose monitor for the first 10 consecutive days during the supplementation period.
  Interventions: Dietary Supplement: Exogenous Ketone Monoester
- Placebo (Placebo Comparator): Participants will consume a flavor-matched placebo drink and undergo the same procedures described in the Experimental Arm
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Exogenous Ketone Monoester — Participants will consume 15g of the oral ketone monoester supplement 15 minutes prior to each meal of the day for 14 days. All meals will be provided throughout the 14-day supplementation period.
  Other Names: KetoneAid KE4 Ketone Ester, D-β-hydroxybutyrate-R 1,3-Butanediol
  Arms: Experimental
Dietary Supplement: Placebo — Participants will consume an equivalent volume (30ml) of the active intervention supplement 15 minutes prior to each meal for 14 days. All meals will be provided throughout the 14-day placebo supplementation period.
  Other Names: Flavor- and volume-matched placebo supplement
  Arms: Placebo

SUMMARY:
Ketone bodies are a fuel source and signaling molecule that are produced by the body during prolonged fasting or if an individuals consistently eats a low-carbohydrate "keto" diet. Blood ketones can be used as a source of energy by the body, but they may also act as signals that impact the functioning of different cells in the body. Recently, the availability of ketone supplements that can be taken orally allows for raising blood ketones without having to fast or eat a "keto" diet. The investigators' studies and those of other researchers have shown that ketone supplementation can lower blood sugar without having to make any other dietary changes. Oral ingestion of ketones may therefore be an effective strategy to improve blood sugar control and influence how cells function.

The main objective of this study is to determine if consuming a ketone supplement 3 times per day (before meals) for 14 days lowers blood sugar and impacts how the body's cells function. The results of this study will be used to guide future recommendations on the utility of ketone supplements for improving health in individuals with, or at elevated risk of, type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Have a type 2 diabetes diagnosis from a physician
* Have stable use of glucose-lowering medications for at least 3 months

Exclusion Criteria:

* Are a competitively trained endurance athlete
* Are actively attempting to gain or lose weight
* Have a history of mental illness or existing neurological disease(s), cardiovascular events (i.e., heart attack, stroke) in the last 2 years
* Have hypoglycemia, irritable bowel syndrome or inflammatory bowel disease
* Are currently using insulin or SGLT2 inhibitors
* Are using more than 2 classes of glucose-lowering medication
* Are currently following a ketogenic diet or taking ketone supplements
* Are unable to commit for a 29-day trial
* Are unable to follow a controlled diet

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Glucose Control: Change in Fructosamine | Day 14 (post-intervention)
  Change in glucose control (from pre-intervention Day 0) will be quantified by serum fructosamine obtained by fasting blood sample in both conditions.

SECONDARY OUTCOMES:
Vascular function | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Vascular function will be assessed by flow mediated dilation of the brachial artery using vascular ultrasound. A cuff will affixed on the forearm, distal to the brachial artery and will be inflated for 5 minutes. Flow mediation dilation will be measured over a 3-minute period following cuff release.
Cognition: N-back test | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Cognition will be assessed using a customized battery of psychometrically validated tests within the domain of executive functions using the computer-based app Inqisit6 Lab (Millisecond). The test will be the n-back test.
Cognition: Digit-symbol substitution test | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Cognition will be assessed using a customized battery of psychometrically validated tests within the domain of executive functions using the computer-based app Inquisit6 Lab (Millisecond). The test will be the digit-symbol substitution test.
Change from baseline plasma insulin at 14 days | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Plasma insulin from venous blood samples will be measured using a high-sensitivity human insulin enzyme-like immunosorbent assay (ELISA) run in duplicate.
Change from baseline plasma free fatty acids at 14 days | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Free fatty acids from venous blood samples will be measured by colorimetric assay run in duplicate.
Change from baseline circulating inflammatory cytokines at 14 days | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Key inflammatory cytokines including CRP will be quantified by Mesoscale Discovery U-PLEX run in duplicate.
Phagocytosis | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Phagocytosis of fluorescent-labelled E. coli by immune cells from whole blood will be quantified by flow cytometry
Oxidative Burst | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  LPS-stimulated oxidative burst by immune cells from whole blood will be quantified by flow cytometry
Degranulation | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Immune cell degranulation will be quantified by enzyme-linked immunosorbent assay run in duplicate (quantifying myeloperoxidase and elastase in whole blood cell culture supernatants).
Immune Cell Phenotyping | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Phenotyping of macrophages and T cells will be quantified by surface and intracellular staining by flow cytometry.
Complete blood count | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  A 5-part white blood cell differential and complete blood count will be quantified by hematology analyzer.
Glycemic Control: 2hr postprandial hyperglycemia | Day 1 through to Day 10
  Glycemic control will be measured by continuous glucose monitoring using the G6 CGM (Dexcom) in both the active and placebo supplement conditions. Glycemic control will be quantified by assessing 2hr postprandial hyperglycemia.
Glycemic Control: 24hr average glucose area under the curve (AUC) | Day 1 through to Day 10
  Glycemic control will be measured by continuous glucose monitoring using the G6 CGM (Dexcom) in both the active and placebo supplement conditions. Glycemic control will be quantified by assessing 24hr average glucose AUC.
Glycemic Control: Fasting glucose | Day 1 through to Day 10
  Glycemic control will be measured by continuous glucose monitoring using the G6 CGM (Dexcom) in both the active and placebo supplement conditions. Glycemic control will be quantified by assessing fasting plasma glucose.
Glycemic Control: Change in Fasting Plasma glucose | Day 14
  Change in fasting plasma glucose (from pre-intervention Day 0) will be measured by fasting blood sample in both the active and placebo supplement conditions.
Glycemic Control: Glycemic variability | Day 1 through to Day 10
  Glycemic control will be measured by continuous glucose monitoring using the G6 CGM (Dexcom) in both the active and placebo supplement conditions. Glycemic control will be quantified by assessing glycemic variability.
Glycemic Control: Time in Target Range | Day 1 through to Day 10
  Glycemic control will be measured by continuous glucose monitoring using the G6 CGM (Dexcom) in both the active and placebo supplement conditions. Glycemic control will be quantified by assessing time in target range.
Glycemic Control: HbA1c | Day 0 (pre-intervention) and Day 14 (post-intervention)
  Glycemic control will be measured by assessing HbA1c using a point-of-care analyzer.
Lipid Panel | Day 0 (pre-intervention) and Day 14 (post-intervention)
  Lipid panel (total cholesterol, high-density cholesterol, low-density cholesterol, triglycerides, non-HDL cholesterol, cholesterol/HDL ratio) will be measured using a point-of-care analyzer.
Body weight | Day 0 (pre-intervention) and Day 14 (post-intervention)
  Change in body weight will be measured using a body weight scale.
Blood pressure | Day 0 (pre-intervention) and Day 14 (post-intervention)
  Change in blood pressure will be measured using an automated blood pressure device. Both systolic and diastolic blood pressure will be measured.
Blood beta-hydroxybutyrate | Day 0 (pre-intervention) and Day 14 (post-intervention)
  Change in fasting blood beta-hydroxybutyrate will be measured using a standard assay.
Physical activity | Day 0 (pre-intervention) to Day 14 (post-intervention)
  Physical activity will be assessed using an accelerometer (activePal) worn throughout the entire intervention period.
Sedentary time | Day 0 (pre-intervention) to Day 14 (post-intervention)
  Sedentary time will be assessed using an accelerometer (activePal) worn throughout the entire intervention period.
Sleeping time | Day 0 (pre-intervention) to Day 14 (post-intervention)
  Sleeping time will be assessed using an accelerometer (activePal) worn throughout the entire intervention period.
Resting heart rate | Day 0 (pre-intervention) and Day 14 (post-intervention)
  Change resting heart rate will be measured using an automated heart rate monitor device.
Waist circumference | Day 0 (pre-intervention) and Day 14 (post-intervention)
  Change in waist circumference will be measures using a measurement tape.

OTHER OUTCOMES:
Supplement acceptability | Day 14
  Acceptability of the supplement (easy of compliance, taste etc.) will be assessed via questionnaire. A 7-point Likert scale will be used.
Hunger and fullness cravings questionnaire | Day 0 (Pre-intervention) through to Day 3
  Perceived hunger will be measured on a visual analogue scale questionnaire assessing hunger and fullness. The questions assessed are:
  1. How hungry do you feel? (0 = I am not hungry at all; 10 = I have never been more hungry)
  2. How satisfied do you feel? (0 = I am completely empty; 10 = I cannot eat another bite)
  3. How full do you feel? (0 = Not at all full; 10 = Totally full)
  4. How much more do you think you can eat? (0 = Nothing at all; 10 = A lot)
T cell Activation | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Markers of T cell activation in whole blood will be quantified by flow cytometry.
Cravings | Day 0 (Pre-intervention) and Day 14 (post-intervention)
  Participants will be asked to report their desire to eat a particular type of food. A visual analogue scale will be used. The questions assessing cravings are:
  1. How often do you experience strong urges to eat particular types of food? (0 = Never; 10 = All the time)
  2. On average how often do you experience a strong urge to eat a particular type of food? (0 = Several times per day; 10 = Once per month)
  3. How strong are these urges you experience to eat particular types of food? (0 = Extremely weak; 10 = Extremely strong)
  4. Are the experiences of strong urges to eat a particular food always of the same strength? (0 = Never; 10 = Always)
  5. How easy is it to ignore this strong urge to eat a particular food? (0 = Very easy; 10 = Impossible)
  6. Is a strong urge to eat a particular food the same as a craving for food? (0 = No; 10 = Yes)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Little, PhD, Principal Investigator — University of British Columbia- Okanagan
Locations (1):
- University of British Columbia Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
The investigators will share individual patient data (de-identified) with researchers upon reasonable request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The de-identified data and associated documents will be made available to researchers upon reasonable request for the duration that is required by the researchers.
Access Criteria: Researchers from accredited institutions will be granted access to the de-identified data and associated documents provided they can show that it will be used for a research-related purpose (e.g., meta-analysis).
URL: http://osf.io

REFERENCES:
- [Derived] Baranowski BJ, Oliveira BF, Falkenhain K, Little JP, Mohammad A, Beaudette SM, Finch MS, Caldwell HG, Neudorf H, MacPherson REK, Walsh JJ. Effect of exogenous beta-hydroxybutyrate on BDNF signaling, cognition, and amyloid precursor protein processing in humans with T2D and insulin-resistant rodents. Am J Physiol Cell Physiol. 2025 Feb 1;328(2):C541-C556. doi: 10.1152/ajpcell.00867.2024. Epub 2025 Jan 13. PMID 39804761